CLINICAL TRIAL: NCT00107731
Title: A Multicenter, Randomized, Parallel-Group, Double-Blind, Phase 3 Comparison of the Efficacy & Safety of Quetiapine Fumarate to Placebo When Used as Adjunct to Mood Stabilizers (Lithium or Valproate) in the Maintenance Treatment of Bipolar I Disorder in Adult Patients (Abbreviated)
Brief Title: Efficacy & Safety of Seroquel Plus Mood Stabilizer in the Maintenance of Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D1447C00126
Record Dates: First submitted 2005-04-07; First posted 2005-04-08 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar I Disorder; Manic Depressive Disorder; Manic Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate; Lithium; Valproic Acid

INTERVENTIONS:
Drug: quetiapine fumarate
Drug: lithium
Drug: divalproex

SUMMARY:
The purpose of this study is to determine whether quetiapine when used as adjunct to lithium or divalproex is safe and effective in the maintenance treatment of adult patients with Bipolar I Disorder. The study consists of enrollment and 2 phases, the Open-label treatment Phase and the Randomized treatment Phase.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Bipolar I Disorder, Most recent episode Manic (296.4x), or Bipolar I Disorder, Most Recent Episode Depressed (296.5x), or Bipolar I Disorder, Most recent Episode Mixed (296.6x), with or without psychotic features, as defined by Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition (DSM-IV)
* At least 1 manic, depressed, or mixed episode in the 2 years prior to the index episode.
* Able to understand and comply with the requirements of the study.

Exclusion Criteria:

* Diagnosis of an anxiety disorder as defined by DSM-IV, which was treated with medication within the past year.
* Known intolerance or lack of response to quetiapine fumarate or to the assigned mood stabilizer, as judged by the investigator.
* Previously randomized into this study or D1447C00126

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710
Dates: Start 2004-04; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of quetiapine versus placebo when used as adjunct therapy to mood stabilizer in increasing time to recurrence of a mood event.

SECONDARY OUTCOMES:
Evaluate the efficacy of quetiapine versus placebo when used as a adjunct therapy to mod stabilizer in increasing time to recurrence of a manic event

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (166):
- United States (36):
  - Research Site, Birmingham, Alabama
  - Research Site, Beverly Hills, California
  - Research Site, Chula Vista, California
  - Research Site, Redlands, California
  - Research Site, San Francisco, California
  - Research Site, Santa Ana, California
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Granite City, Illinois
  - Research Site, Libertyville, Illinois
  - Research Site, Schaumburg, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Metairie, Louisiana
  - Research Site, Glen Burnie, Maryland
  - Research Site, Kalamazoo, Michigan
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Brooklyn, New York
  - Research Site, Olean, New York
  - Research Site, Rochester, New York
  - Research Site, Morganton, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Havertown, Pennsylvania
  - Research Site, Media, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Conroe, Texas
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin
- Australia (9):
  - Research Site, Greenwich, New South Wales
  - Research Site, Brisbane, Queensland
  - Research Site, Everton Park, Queensland
  - Research Site, Southport, Queensland
  - Research Site, Glenside, South Australia
  - Research Site, Box Hill, Victoria
  - Research Site, Dandenong, Victoria
  - Research Site, Epping, Victoria
  - Research Site, Richmond, Victoria
- Belgium (7):
  - Research Site, Assebroek
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Kortenberg
  - Research Site, Manage
  - Research Site, St-Denijs-Westrem
  - Research Site, Waregem
- Bulgaria (4):
  - Research Site, Kardzhali
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Czechia (5):
  - Research Site, Jeseník
  - Research Site, Litomolice
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Pterova
- Finland (5):
  - Research Site, Espoo
  - Research Site, Harjavalta
  - Research Site, Helsinki
  - Research Site, Kellokoski
  - Research Site, Seinäjoki
- France (9):
  - Research Site, Besançon
  - Research Site, Bourg-en-Bresse
  - Research Site, La Rochelle
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (8):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Heidelberg
  - Research Site, Homburg
  - Research Site, München
  - Research Site, Regensburg
  - Research Site, Saarbrücken
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Füzesabony
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Kistarcsa
  - Research Site, Pécs
- Italy (15):
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Brescia
  - Research Site, Cagliari
  - Research Site, Civitanova Marche
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, La Spezia
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Siena
  - Research Site, Trieste
- Norway (7):
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Bryne
  - Research Site, Namsos
  - Research Site, Oslo
  - Research Site, Ottestad
  - Research Site, Skien
- Poland (17):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Choroszcz
  - Research Site, Gdansk
  - Research Site, Gorlice
  - Research Site, Janów Lubelski
  - Research Site, Krakow
  - Research Site, Lipno
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Nowy Targ
  - Research Site, Poznan
  - Research Site, Starogard Gdański
  - Research Site, Szczecin
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Zubki
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Saratov
- South Africa (5):
  - Research Site, Bloemfontein
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Krugersdorp
  - Research Site, Pretoria
- Spain (13):
  - Research Site, Barcelona, Barcelona
  - Research Site, Terrassa, Barcelona
  - Research Site, Puerto Real, Cádiz
  - Research Site, Granada, Granada
  - Research Site, Madrid, Madrid
  - Research Site, Oviedo, Oviedo
  - Research Site, Langreo, Principality of Asturias
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Seville, Sevilla
  - Research Site, Bilbao
  - Research Site, Guadalajara
  - Research Site, Santiago de Compostela
  - Research Site, Vigo
- Sweden (6):
  - Research Site, Falköping
  - Research Site, Linköping
  - Research Site, Ludvika
  - Research Site, Sollentuna
  - Research Site, Stockholm
  - Research Site, Sundsvall
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
- United Kingdom (7):
  - Research Site, Birmingham
  - Research Site, London
  - Research Site, Oxford
  - Research Site, Runcorn
  - Research Site, Ryhope
  - Research Site, Surbiton
  - Research Site, Welwyn Garden City

REFERENCES:
- [Derived] Suppes T, Vieta E, Gustafsson U, Ekholm B. Maintenance treatment with quetiapine when combined with either lithium or divalproex in bipolar I disorder: analysis of two large randomized, placebo-controlled trials. Depress Anxiety. 2013 Nov;30(11):1089-98. doi: 10.1002/da.22136. Epub 2013 Jun 12. PMID 23761037